CLINICAL TRIAL: NCT05702099
Title: Effect of Simultaneous Cystectomy on Ovarian Reserve in Cases of Adnexal Detorsion
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Evrim Ebru Kovalak, Principal investigator, Doctor, Gynecology and obstetrics specialist, Bagcilar Training and Research Hospital
Other Study IDs: GOKAEK/2017-577
Record Dates: First submitted 2022-12-21; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Torsion
Keywords: ovarian torsion; cystectomy; ovarian reserve
MeSH Terms: conditions — Ovarian Torsion | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Detorsion: The group in which only adnexal detorsion was performed during the operation (Because there is no ovarian mass)
  Interventions: Diagnostic Test: ultrasonography
- Detorsion+cystectomy: Women with an ovarian mass who underwent emergency surgery for torsion, who underwent both detorsion and cystectomy in the same session.
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — By performing transvaginal or transabdominal ultrasonography on women, ovarian volume will be calculated and antral follicle will be counted.

SUMMARY:
There are mostly ovarian cysts under adnexal torsion from gynecological emergencies. There are many studies in the literature examining the effect of adnexal detorsion on ovarian reserve. However, there is no study in the literature examining the effect of concomitant cystectomy. In this study, the investigators aimed to investigate whether the cystectomy procedure performed together with detorsion has an additional effect on the ovarian reserve in cases of ovarian torsion with cysts.

DETAILED DESCRIPTION:
All women who underwent emergency surgery in the investigators' obstetrics and gynecology department since April 2015 due to adnexal torsion were analyzed. All patients who underwent ovarian detorsion (Group 1) and ovarian detorsion+cystectomy (Group 2) were called for control between 6-12 months postoperatively. In all patients, the sizes of both ovaries and the number of antral follicles were counted by ultrasonography by 2 physicians who did not know the detorsion side beforehand. All women will be compared within and between groups in terms of ovarian sizes and antral follicle numbers.

ELIGIBILITY:
Inclusion Criteria:

* All women who underwent emergency surgery for ovarian torsion

Exclusion Criteria:

* Those who underwent oophorectomy with suspicion of malignancy
* When faced with spontaneously amputated ovary due to chronic or acute torsion
* Women with only salpinx torsion

Ages: 15 Years to 63 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All women between the ages of 15-63 who underwent emergency surgery for ovarian torsion.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Ovarian volume difference between groups | postoperative 6-12 months
  To analyze whether there is a difference between the ovarian reserve parameters of women who underwent detorsion and detorsion+cystectomy. With ultrasonographic imaging, both ovaries will be evaluated for ovarian volume ( V = length × width × height × π/6) (cm3). Both the affected ovary will be compared with the contralateral ovary and the affected ovaries will be compared between groups.
The number of antral follicles difference between groups | postoperative 6-12 months
  To analyze whether there is a difference between the ovarian reserve parameters of women who underwent detorsion and detorsion+cystectomy. With ultrasonographic imaging, both ovaries will be evaluated for the number of antral follicles. Both the affected ovary will be compared with the contralateral ovary and the affected ovaries will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Ebru Kovalak, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Teaching and Research Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bozdag G, Demir B, Calis PT, Zengin D, Dilbaz B. The impact of adnexal torsion on antral follicle count when compared with contralateral ovary. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):632-5. doi: 10.1016/j.jmig.2014.01.007. Epub 2014 Jan 21. PMID 24462592
- [Result] Calis P, Bozdag G, Karakoc Sokmensuer L, Kender N. Does ischemia-reperfusion injury affect ovarian reserve and follicle viability in a rat model with adnexal torsion? Eur J Obstet Gynecol Reprod Biol. 2015 Feb;185:126-30. doi: 10.1016/j.ejogrb.2014.12.006. Epub 2014 Dec 23. PMID 25575140